CLINICAL TRIAL: NCT05398575
Title: Music Listening for Cardiorespiratory Exercise in Inpatient Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other); Regionshospital Nordjylland (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Music cardio stroke
Record Dates: First submitted 2022-04-19; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment with tailored music playlist (Experimental): Music playlist tailored for a group of 5-8 individuals.
  Interventions: Behavioral: Music
- Standard treatment with radio music (Active Comparator): Listening to local radio channel with music
  Interventions: Behavioral: Music
- Standard treatment without music (No Intervention): Standard physiotherapy with no audio intervention

INTERVENTIONS:
Behavioral: Music — Participants listen to music during physiotherapy rehabilitation (tailored or radio music)
  Arms: Standard treatment with radio music; Standard treatment with tailored music playlist

SUMMARY:
Stroke survivors struggle to meet clinical recommendations for physical exercise duration and intensity. During the past two decades, music interventions have increasingly shown effectiveness in several motor tasks in stroke rehabilitation. Additionally, music has been found effective in increasing exercise performance in athletes and other clinical populations. Based on a meta-theoretical review paper by Clark, Baker & Taylor (2016), it was hypothesized that the therapeutic effects of music in physical exercise is modulated by the preference and task-specificity of the music. We will test this hypothesis using a three-armed randomized cross-over design comprised of the following auditory conditions: 1) a group-tailored playlist 2) radio as active control and 3) a non-music control condition during cycle ergometry cardiorespiratory exercise sessions. Participants are inpatient stroke survivors undergoing rehabilitation between 2-12 weeks post infarct.

ELIGIBILITY:
Inclusion Criteria:

* between 2-12 weeks post ischemic or hemorrhagic stroke
* assessed eligible to participate in cardiorespiratory exercise by the patient's primary physiotherapist and interdisciplinary team -≥18 years old

Exclusion Criteria:

* uncontrolled medical contraindications for physical activity
* severe hearing deficit or cochlear implants
* severe deficit of both auditory and visual communication not allowing for guiding the patient in the exercise task

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Heart rate reserve | Proportion of time during the 30 minutes session
  Time spent in therapeutic heart rate zone
Exercise time | Proportion of time during the 30 minutes session
  Time spent actively participating in the physiotherapy session

SECONDARY OUTCOMES:
Feeling scale | Immediately before and after the intervention.
  11 point Likert scale rating affective valence (current feeling state)
Evaluation of condition | Immediately after the intervention
  Rating of preferred audio condition on a 10 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Mazhari-Jensen, MA, Principal Investigator — Aalborg University
Locations (1):
- North Denmark Region, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No